CLINICAL TRIAL: NCT02853357
Title: Short-term Effects of Thoracic Spine Thrust Manipulation for Individuals With Low Back Pain: A Randomized Control Trial
Brief Title: Thoracic Spine Manipulation for Individuals With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Rocky Mountain University of Health Professions (Other)
Responsible Party: Principal Investigator, Laura Fisher, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00105566
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain
Keywords: Thoracic manipulation; Low back pain; Core strengthening; Thoracic spine thrust manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): The control group includes randomized participants that will receive a sham manipulation. Participants will also complete the standard set of core strengthening exercises.
  Interventions: Other: Sham Manipulation; Other: Core Strengthening Exercises
- Manipulation (Experimental): The manipulation group includes randomized participants that will receive a thoracic spine thrust manipulation. Participants will also complete the standard set of core strengthening exercises.
  Interventions: Other: Manipulation; Other: Core Strengthening Exercises

INTERVENTIONS:
Other: Manipulation — Middle Thoracic: Participants are placed in the supine position with their arms over their chest. The clinician rolls the participant to their side and places the fulcrum at the desired thoracic segment and the participant is rolled back onto the clinician's hand. The participant is instructed to take a deep breath. As the participant is exhaling, the clinician uses his body to push through the participant's arms to perform a high velocity thrust in an anterior to posterior directed force. Lower Thoracic: With the patient in a prone position, the clinician achieves a "skin lock" with both pisiforms over the transverse processes of the target vertebra. The clinician then uses his body to push down through his arms to perform a high-velocity, low-amplitude posterior to anterior thrust.
  Other Names: Thoracic Manipulation; Thoracic spine thrust manipulation; Lower thoracic manipulation; Middle thoracic manipulation
  Arms: Manipulation
Other: Sham Manipulation — The participants are positioned in prone and the clinician's hands are placed with the pisiforms of each hand over the transverse processes of the target vertebra. The clinician will only apply minimal pressure and slide the hands across the skin to mimic the manipulative thrust. This sham procedure has been shown to be an adequate sham comparator for spinal manipulative therapy (SMT) with similar expectations and believability as SMT active treatment
  Other Names: Sham thoracic manipulation
  Arms: Control
Other: Core Strengthening Exercises — Both groups will receive the following exercises at each visit. The core strengthening (core strengthening) exercises are a standard protocol used by Richardson et al and Franca et al which are proposed to target muscles responsible for segmental stabilization, specifically the transverse abdominis (TrA) and the lumbar multifidi (LM). Exercises will include: TrA exercises in 4 point kneeling and in supine with flexed knee, LM exercises in prone, and co-contraction of TrA and LM in upright position. Three sets of 15 repetitions will be done for each exercise.
  Other Names: Transverse Abdominis exercises; Lumbar Multifidi exercises

SUMMARY:
The purpose of this study is to determine the short-term effects of thoracic spine thrust manipulation on participants with low back pain. Participants in this study will be randomized to receive either the lower thoracic spinal manipulation and a standard set of exercises, or a sham manipulation and the same standard set of exercises. It is hypothesized that thoracic manipulation when combined with core strengthening exercises will have positive short term improvements in pain and function for patients with LBP as compared to a sham manipulation combined with core strengthening exercises.

DETAILED DESCRIPTION:
This study aims to use a randomized controlled trial design to investigate the effects of thoracic spinal manipulation in conjunction with core strengthening exercises when compared to a sham manipulation and core strengthening exercises on patients with low back pain. Core strengthening exercises have been shown to improve pain and functional status in patients with non-specific low back pain when compared to conventional exercise. However, there is strong evidence to suggest that exercise alone is not adequate for the management of low back pain. Spinal manipulation has demonstrated promising results for the management of low back pain, but it is unclear whether the targeted location of manipulation is important. It is hypothesized that thoracic manipulation when combined with core strengthening exercises will have positive short term improvements in pain and function for patients with LBP as compared to a sham manipulation combined with core strengthening exercises based on the theory of regional interdependence. The specific aims of the study are as follows:

1. To determine the effects of thoracic spine manipulation and core strengthening exercise on function in individuals with low back pain, specifically measured by changes in Modified Oswestry Low Back Pain Disability Questionnaire (MODQ).
2. To determine the participant's perception of improvement following thoracic spine manipulation and core exercises, measured by global rating of change (GROC), when compared to a sham manipulation.
3. To determine the effects of thoracic spine manipulation and core exercises on fear avoidance, measured by fear-avoidance belief questionnaire (FABQ), on individuals with low back pain.
4. To determine the effects of thoracic spine manipulation and core exercises on pain using numeric pain rating scale (NPRS).

The ability to demonstrate the effectiveness of a manipulation targeted at the thoracic spine in conjunction with core exercises could provide clinicians a simple, effective treatment strategy for low back pain that not only has minimal injury risk, but has the potential to improve pain and function, ultimately decreasing the healthcare costs associated with low back pain.

The effects of treatment on disability, fear-avoidance, and pain will be analyzed using a 2x2 repeated measures multivariate analysis of variance (MANCOVA), with pre/post-test measures and time as the two factors and duration of symptoms serving as a covariate. An independent t test will be used to determine differences for the Global Rating of Change between groups at follow up, and the number needed to treat (NNT) will be calculated. Spinal manipulation has some potentially serious risks including, fracture, numbness, tingling, or injury to the spinal cord. However, these risks are very low in the thoracic spine where manipulation is targeted during this study. In a recent systematic review which evaluated the safety of thoracic spine manipulation, the authors found only seven cases of serious trauma which have resulted from thoracic spine manipulation. The majority of these cases were performed by a chiropractor and it is unsure whether participants had contraindications to manipulation. In order to mitigate these risks, participants will be thoroughly screened for contraindications to spinal manipulation. If an adverse event does occur, the participant will be referred to the appropriate provider and their participation in the study will be discontinued.

ELIGIBILITY:
The precise inclusion criteria scores are not indicated in the inclusion criteria below to avoid inappropriate self-selection of participants. After enrollment and data collection are complete, the investigators will list the actual minimum scores allowable for inclusion, when the data can no longer be skewed.

Inclusion Criteria:

* A certain minimum pain intensity score on an 11-point numeric pain rating scale (ranging from 0-10 points)
* A certain minimum disability rain on the Modified Oswestry Disability Questionnaire
* Individuals who have received a prescription for physical therapy for low back pain

Exclusion Criteria:

* Contraindications to spinal manipulation such as osteoporosis, active cancer, previous spinal surgery, spinal fracture, acute rheumatic disease, active tuberculosis, pregnancy, active infections of the vertebra or intervertebral disc, any neurological evidence suggesting compromise of the nerve roots or spinal cord (changes in myotomal strength, deep tendon reflexes, or sensation), or cauda equina syndrome
* Insufficient English skills to complete questionnaires
* Are involved in litigation or a workman's compensation claim

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Modified Oswestry Disability Questionnaire (MODQ) | Administered at the initial and final sessions (no more than 2 weeks apart)
  The MODQ is a functional scale assessing the impact of low back pain on daily activities by assigning a disability score according to the answered questions. The scale includes 10 questions regard the level of pain and interference with several physical activities including: sleeping, lifting, travelling, self-care, and social life. Each question has six possible responses (scored from 0 to 5), and patients are asked to pick the one that most accurately responds to their condition. The sum of the response is divided by the total possible score and multiplied by 100 to receive a percentage of disability with 0% corresponding to no disability and 100% corresponding to a great deal of disability.

SECONDARY OUTCOMES:
Change from Baseline on Numeric Pain Rating Scale (NPRS) | Administered at the initial and final sessions (no more than 2 weeks apart)
  An 11-point numeric pain rating scale will be used to assess pain before and after treatment. The scale ranges from 0 "no pain" to 10 "worst possible pain."
Change from Baseline on Numeric Pain Rating Scale (NPRS) | Administered at the initial session and 3 months after the final session
  An 11-point numeric pain rating scale will be used to assess pain before and after treatment. The scale ranges from 0 "no pain" to 10 "worst possible pain."
Change from Baseline on Fear-Avoidance Belief Questionnaire (FABQ) | Administered at the initial and final sessions (no more than 2 weeks apart)
  The FABQ is used to quantify individual's fear avoidance beliefs and LBP specifically regarding avoiding activity. The FABQ is divided into physical activity (FABQ-PA) and work subscales (FABQ-W) in which patients rate their agreement of each statement on a seven point Likert scale (0 is completely disagree and 6 is completely agree).
Change from Baseline on Fear-Avoidance Belief Questionnaire (FABQ) | Administered at the initial session and 3 months after the final session
  The FABQ is used to quantify individual's fear avoidance beliefs and LBP specifically regarding avoiding activity. The FABQ is divided into physical activity (FABQ-PA) and work subscales (FABQ-W) in which patients rate their agreement of each statement on a seven point Likert scale (0 is completely disagree and 6 is completely agree).
Global Rating of Change Scale (GROC) | Administered at the final session (no more than 2 weeks after the initial evaluation)
  The GROC is used to assess self-perceived improvement of the intervention. The GROC is a 15-point scale ranging from -7 (a very great deal worse) to 0 (about the same) to +7 (a very great deal better).
Change on the Global Rating of Change Scale (GROC) | Administered at the final session (no more than 2 weeks after the initial evaluation) and 3 months after the final session
  The GROC is used to assess self-perceived improvement of the intervention. The GROC is a 15-point scale ranging from -7 (a very great deal worse) to 0 (about the same) to +7 (a very great deal better).
Change from Baseline on Modified Oswestry Disability Questionnaire (MODQ) | Administered at the initial session and 3 months after the final session
  The MODQ is a functional scale assessing the impact of low back pain on daily activities by assigning a disability score according to the answered questions. The scale includes 10 questions regard the level of pain and interference with several physical activities including: sleeping, lifting, travelling, self-care, and social life. Each question has six possible responses (scored from 0 to 5), and patients are asked to pick the one that most accurately responds to their condition. The sum of the response is divided by the total possible score and multiplied by 100 to receive a percentage of disability with 0% corresponding to no disability and 100% corresponding to a great deal of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Fisher, BS, DPT, OCS, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inani SB, Selkar SP. Effect of core stabilization exercises versus conventional exercises on pain and functional status in patients with non-specific low back pain: a randomized clinical trial. J Back Musculoskelet Rehabil. 2013;26(1):37-43. doi: 10.3233/BMR-2012-0348. PMID 23411647
- [Background] Smith BE, Littlewood C, May S. An update of stabilisation exercises for low back pain: a systematic review with meta-analysis. BMC Musculoskelet Disord. 2014 Dec 9;15:416. doi: 10.1186/1471-2474-15-416. PMID 25488399
- [Background] Mintken PE, Cleland JA, Carpenter KJ, Bieniek ML, Keirns M, Whitman JM. Some factors predict successful short-term outcomes in individuals with shoulder pain receiving cervicothoracic manipulation: a single-arm trial. Phys Ther. 2010 Jan;90(1):26-42. doi: 10.2522/ptj.20090095. Epub 2009 Dec 3. PMID 19959652
- [Background] Michener LA, Kardouni JR, Lopes Albers AD, Ely JM. Development of a sham comparator for thoracic spinal manipulative therapy for use with shoulder disorders. Man Ther. 2013 Feb;18(1):60-4. doi: 10.1016/j.math.2012.07.003. Epub 2012 Aug 9. PMID 22883130
- [Background] Richardson C, Hodges P, Hides J. Therapeutic exercise for lumbopelvic stabilization. Churchill Livingstone London; 2004.
- [Background] Richardson CA, Jull G, Hodges P, Hides J. Therapeutic exercise for spinal segmental stabilization in low back pain: scientific basis and clinical approach. Churchill Livingstone; 1999.
- [Result] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Result] de Oliveira RF, Liebano RE, Costa Lda C, Rissato LL, Costa LO. Immediate effects of region-specific and non-region-specific spinal manipulative therapy in patients with chronic low back pain: a randomized controlled trial. Phys Ther. 2013 Jun;93(6):748-56. doi: 10.2522/ptj.20120256. Epub 2013 Feb 21. PMID 23431209
- [Result] Masaracchio M, Cleland JA, Hellman M, Hagins M. Short-term combined effects of thoracic spine thrust manipulation and cervical spine nonthrust manipulation in individuals with mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2013 Mar;43(3):118-27. doi: 10.2519/jospt.2013.4221. Epub 2012 Dec 7. PMID 23221367
- [Result] Franca FR, Burke TN, Hanada ES, Marques AP. Segmental stabilization and muscular strengthening in chronic low back pain: a comparative study. Clinics (Sao Paulo). 2010;65(10):1013-7. doi: 10.1590/s1807-59322010001000015. PMID 21120303
- [Result] Maughan EF, Lewis JS. Outcome measures in chronic low back pain. Eur Spine J. 2010 Sep;19(9):1484-94. doi: 10.1007/s00586-010-1353-6. Epub 2010 Apr 17. PMID 20397032